CLINICAL TRIAL: NCT06746922
Title: The Effect of Intermittent Theta Burst Stimulation to the Primary Motor Cortex on Pain Intensity, Pain Catastrophizing, Quality of Life and Mood in Fibromyalgia Patients
Brief Title: Intermittent Theta Burst Stimulation in Fibromyalgia Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ayhan Aşkın, MD, Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-KAEK-23
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia; Transcranial Magnetic Stimulation Repetitive; Pain
Keywords: Fibromyalgia; intermittent theta burst stimulation; pain; Pain Catastrophizing; Revised Fibromyalgia Impact Questionnaire; Hospital Anxiety and Depression Scale
MeSH Terms: conditions — Fibromyalgia; Pain; Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation group (Experimental): Patients will receive intermittent theta burst stimulation (iTBS) to the primary motor cortex, one session per day for a total of 10 sessions.
  Interventions: Device: Intermittent theta-burst stimulation
- Sham stimulation group (Sham Comparator): Patients will receive sham treatment for one session per day for a total of 10 sessions.
  Interventions: Device: Sham Intermittent theta-burst stimulation

INTERVENTIONS:
Device: Intermittent theta-burst stimulation — Neuro-MS/D (Neurosoft) rTMS device will be used for stimulation with an angulated figure-of-eight coil. Neuronavigation system will be used to determine the application site. Before each session, active motor threshold (aMT) will be determined by obtaining a motor evoked potential with an amplitude of >200μV in the EMG recording of the first dorsal interosseous muscle (FDI), which is slightly contracted (10-20% of maximum contraction) in at least five out of 10 stimuli delivered to the primary motor cortex. The handle will be held at a 45° angle to the sagittal plane, pointing backwards and laterally to create posterior-anterior current flow in the brain. The stimulation parameters are as follows:
  Parameters:
  Stimulation type:Burst Stimulus amplitude (% MT): 80 Burst frequency in sequence (Hz):5 Pulse frequency within burst (Hz):50 Number of bursts in the sequence: 10 Number of series:20 Interval between sequences: 8 sec Total time: 3min 47sec Total number of pulses: 600
  Arms: Active stimulation group
Device: Sham Intermittent theta-burst stimulation — In the sham application, the probe of the transcranial magnetic stimulation device will be placed in the vertical position and held perpendicular to the vertex and applied at an ineffective dose so that the patient hears the same sound. In order for the device to produce the same sound and warning sounds as the active application, it will be operated at the lowest operating power of 1 power. In the device operating at this power, there is no possibility of any warning due to the upright position of the probe.
  Arms: Sham stimulation group

SUMMARY:
Research on repetitive transcranial magnetic stimulation therapy in fibromyalgia syndrome (FMS) is increasing rapidly. High-frequency rTMS administration to FMS patients is reported to restore intracortical facilitation and provide successful pain relief. This finding supports restoration of cortical stimulation as one of the possible mechanisms of action for rTMS. One treatment protocol is intermittent theta burst stimulation (iTBS, a variant of excitatory rTMS). Although there are many treatment protocols, there are few widely accepted treatment schemes in the literature. In fibromyalgia syndrome, there is no study in the literature. It was planned to include at least 30 patients aged 18-65 years who were admitted to İzmir Katip Çelebi University Atatürk Training and Research Hospital Physical Medicine and Rehabilitation Outpatient Clinic or hospitalized in the ward and diagnosed with fibromyalgia syndrome according to the 2016 criteria. This study has a prospective, parallel group, randomized, sham-controlled study design. A total of 30 fibromyalgia patients will be randomized into 2 groups and will receive a total of 10 sessions of transcranial magnetic stimulation to the primary motor cortex with intermittent theta bust stimulation technique or sham application. Patients will continue their current fibromyalgia treatment.Numeric Rating Scale-pain intensity (NRS-pain), revised Fibromyalgia Impact Questionnaire (FIQR), Pain Catastrophizing Scale (PCS), Hospital Depression Anxiety Scale (HADS) will be used in the evaluation of the patients.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is a chronic condition characterized by generalized body pain, fatigue, sleep disturbance, impaired cognitive function and anxiety of unknown etiology. Potential causes include genetic, neurologic, psychological, sleep and immunologic factors. In the literature, complaints or symptoms reported by more than 25% of patients with FMS include widespread body pain, fatigue, morning stiffness, headache, paresthesia, sleep disturbance, subjective swelling, dry mouth, irritable bowel, dysmenorrhea, joint hypermobility, temporomandibular joint dysfunction, dermographism, Raynaud's phenomenon and reticular skin discoloration. Although some factors are known to predispose individuals to FMS (e.g. genes, adverse life events and physical trauma), the etiology of FMS is still unknown.

One of the best-supported hypotheses regarding its pathophysiology is the presence of central sensitization to pain and deficiencies in endogenous pain inhibitory mechanisms. Its prevalence has been reported as 0.2% to 6.6%. This rate increases to 2.4% to 6.8% in women. This rate increases in the 40-60 age group and in Turkey, the prevalence of fibromyalgia is reported to be 3.6% in women, with the highest rate (10.1%) observed in women aged 50-59 years. Studies show that fibromyalgia is more common in the female gender, among people with low education and socioeconomic status, and in the 40-60 age group.

The clinical picture of the patients shows that the pain is usually localized at first, but then involves many muscle groups. Hyperalgesia and allodynia are important features of fibromyalgia, although it can often be described as burning, gnawing pain, stiffness or aching sensation. Patients often complain of swollen joints and paresthesia despite the absence of any objective clinical findings during physical examination. Pain is often exacerbated by cold and damp weather, inadequate sleep, physical and mental stress.

There is no gold standard for the diagnosis of fibromyalgia. There are no laboratory markers or tests for the diagnosis of FMS and the diagnosis is made entirely clinically. Although the 1990 and 2010 criteria were also used in the diagnosis of FMS until recently, the latest version of the 2016 American College of Rheumatology (ACR) revised criteria are used. According to the 2016 ACR diagnostic criteria, the presence of generalized pain defined as pain in at least four of the five regions (four quadrants and axial) (however, jaw, chest, abdomen, headache and facial pain should not be included in the quadrant or regional definition of generalized pain), symptoms should be present at a similar level for at least 3 months, and scores should be WPI ≥ 7 and SS ≥ 5 or WPI 4-6 and SS ≥ 9.

The main goal of treatment should be to alleviate the patient's symptoms and improve quality of life. Current evidence-based guidelines emphasize the value of multimodal therapies, including both non-pharmacological and selected pharmacological treatments tailored to individual symptoms, including pain, fatigue, sleep problems and mood problems.According to EULAR, in the treatment of fibromyalgia, non-pharmacological treatment should be the first-line treatment and, if there is a lack of efficacy, individualized treatment should be applied, which may include pharmacological treatment according to the patient's needs, and these recommendations are now firmly evidence-based. Through various interventions such as non-pharmacological treatment methods; cognitive-behavioral therapy (CBT), physical therapy, mindfulness, acupuncture, physical therapy and exercise, mindfulness and meditation, acupuncture and acupressure, individuals can develop effective strategies to cope with pain, improve their functional abilities and increase their quality of life. Exercise has been shown to reduce stress, depression and anxiety and has been successfully applied in the treatment of chronic pain disorders such as chronic pelvic pain, migraine and fibromyalgia. There are different mechanisms that may explain the beneficial effect of exercise on fibromyalgia, including causing an increase in endogenous opioids, stimulating brain structures involved in diminished analgesic pathways and/or maintaining the balance between excitatory (glutamate) and inhibitory (GABA) neurotransmitters in the brain. It has been shown that the greatest improvement in fibromyalgia patients is seen after prolonged (12 weeks) moderate intensity aerobic training. Another form of non-pharmacological treatment is Cognitive Behavioral Therapy, which involves educating patients about their pain, how to cope with their pain, such as relaxation training, and how to apply these cognitive coping techniques in real life situations. Among recent studies on fibromyalgia treatment, EEG-guided neurofeedback targeting specific brain regions such as the anterior cingulate cortex and supplementary motor area has shown initial success in alleviating chronic pain in fibromyalgia patients.

A recent study has shown that stimulation of the left DLPFC with repetitive transcranial magnetic stimulation (rTMS) has a role in pain management and physical role functioning, and that it affects the activity of a network of structures involved in the integration and modulation of pain signals, including the thalamus as a mechanism. Non-invasive brain stimulation is increasingly recommended as a treatment for a variety of neurological and psychiatric disorders, including pain, depression, anxiety and compulsive disorders.

Among pharmacologic treatments, duloxetine, a balanced serotonin and norepinephrine dual reuptake inhibitor, is first in line. Drugs that inhibit the reuptake of serotonin and norepinephrine potentiate monoamine neurotransmission along oppressive descending pathways in the spinal cord, thereby reducing nociceptive afferent transmission in ascending spinal pain pathways. The effect of drugs such as duloxetine is independent of their effect on depression, with the onset of benefit occurring within days, earlier and at lower doses than in depression. Common side effects include nausea, headache, dry mouth, insomnia, constipation, dizziness, fatigue, somnolence, excessive sweating and diarrhea. Another therapeutic agent is amitriptyline, but its side effect profile is higher than that of other agents, so its use has been less common, although randomized placebo-controlled clinical trials have shown the efficacy of amitriptyline in the treatment of painful conditions, including fibromyalgia and neuropathies, such as postherpetic, diabetic or chemotherapy-associated neuropathies and chronic arm pain. Another therapeutic agent is pregabalin, approved by the FDA for the relief of neuropathic pain associated with fibromyalgia as well as diabetic peripheral neuropathy, spinal cord injury and postherpetic neuralgia. The recommended therapeutic dosage for FMS is 300mg to 450mg daily, with an initial dose of 150mg/day divided into two daily doses. The dosage can be increased to 300mg per day within 1 week of starting treatment. In patients whose pain is not optimally relieved with 300 mg/day, the dosage can be increased to 450 mg/day divided into two daily doses. In a randomized, double-blind, flexible-dose study with gabapentin, it was shown to significantly reduce fibromyalgia-related pain as measured by the BPI mean pain intensity score, the primary efficacy measure, compared with placebo (1200-2400 mg daily).

Especially when rTMS studies are considered, different rTMS treatment protocols have been reported in fibromyalgia patients in previous studies. There are sham-controlled studies in which primary motor cortex and dorsolateral prefrontal cortex were stimulated. Tekin et al. reported that 10hz rTMS treatment applied to the primary motor cortex was effective in decreasing global pain scores and increasing quality of life. Short et al. investigated the effect of 10hz rTMS application to the left dorsolateral prefrontal cortex (DLPFC) on pain, quality of life, depression and anxiety in a randomized controlled study. That study supported the hypothesis that high frequency rTMS applied to the left DLPFC may reduce fibromyalgia pain as an adjunct to pharmacotherapy. A recent network meta-analysis revealed that treatment using 20Hz rTMS was the optimal stimulation frequency for reducing chronic pain. While lower frequencies have also shown significant pain reduction, it has been reported that the effects dissipate over time. In another network meta-analysis investigating the efficacy of different types of neuromodulation on fibromyalgia, it was reported that high frequency rTMS on the primary motor cortex showed significant efficacy on pain and functionality. In the 2024 update of a meta-analysis evaluating the effect of rTMS applied to the DLPFC on pain, it was reported that DLPFC-rTMS had no effect on neuropathic pain, although it had potential benefits for the negative emotions of chronic pain with the inclusion of recent large-sample studies.When this study was planned, there was no research on the effect of intermittent theta burst stimulation applied to the primary motor cortex on the disease course in FMS patients. Although intermittent theta burst stimulation is a known application technique with high-frequency activation potential, it is not yet clear how it will affect FMS patients.

The aim of this study was to determine the efficacy of intermittent theta burst stimulation to the primary motor cortex on pain intensity, pain catastrophizing, quality of life and mood in FMS patients.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Being diagnosed with fibromyalgia syndrome (according to 2016 criteria)
* Average pain intensity of NRS ≥ 4/10
* Fibromyalgia treatment was stable for the last 3 months and no treatment change was planned during the study

Exclusion Criteria:

* Having a clinical condition that would constitute a contraindication for TMS (metallic implant, cardiac pacing, pregnancy, epilepsy, head trauma, history of cranial operation...)
* Presence of malignancy
* Systemic rheumatologic diseases
* Major orthopedic problems limiting activities of daily living (gait disturbance or fracture sequelae limiting joint mobility, prostheses, nerve-tendon injuries)
* Serious neurological diseases (increased intracranial pressure, presence of space-occupying lesions in the brain, history of epilepsy, presence of cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, history of previous head trauma causing loss of consciousness)
* Alcohol or drug addiction
* History of major depression/personality disorder or psychosis
* Having received TMS treatment before
* Taking benzodiazepine, gabapentin/pregabalin or anticonvulsant medications that have the potential to interfere with intermittent theta burst stimulation treatment or have taken them within the last 4 weeks
* Pregnant or planning pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Numeric Rating Scale | (1) at the beginning of the treatment (T0), (2) at the 1st week (T1), (3) at the 2nd week (T2), (4) four weeks after the end of the treatment (T3).
  The numeric rating scale for pain that is a unidimensional measure of pain intensity in adults, including those with chronic pain.The common format is a horizontal bar or line. Similar to the visual analog scale, the numeric rating scale for pain is anchored by terms describing pain severity extremes. The 11-point numeric scale ranges from 0 representing one pain extreme (e.g. "no pain") to 11 representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
Change from baseline in the Revised Fibromyalgia Impact Questionnaire | (1) at the beginning of the treatment (T0), (2) at the 2nd week (T2), (3) four weeks after the end of the treatment (T3).
  The Revised Fibromyalgia Impact Questionnaire (FIQR) has 21 individual questions. All questions are based on an 11-point numeric rating scale of 0 to 10, with 10 being 'worst'. As in the FIQ, all questions are framed in the context of the past 7 days. Following the convention used in the FIQ, the FIQR is divided into three linked sets of domains: (a) 'function' (contains 9 questions versus 11 in the FIQ), (b) 'overall impact' (contains 2 questions, as in the FIQ) but the questions now relate to the overall impact of FM on functioning and the overall impact symptom severity, and (c) 'symptoms' (contains 10 questions versus 7 in the FIQ)
Change from baseline in the Pain Catastrophizing Scale | (1) at the beginning of the treatment (T0), (2) at the 2nd week (T2), (3) four weeks after the end of the treatment (T3).
  The Pain Catastrophizing Scale (PCS) is a 13-item self-report measure designed to assess catastrophic thinking related to pain among adults with or without chronic pain.13 items rated on 5-point Likert scales, from (0) not at all to (4) all the time. Higher score indicates higher level of catastrophizing.
  Item scores are summed into a total score (PCS-T) and three subscale scores:
  * Rumination (PCS-R): Items 8, 9, 10, and 11
  * Magnification (PCS-M): Items 6, 7, 13
  * Helplessness (PCS-H): Items 1, 2, 3, 4, 5, and 12 Minimum total score = 0, maximum total score = 52 Subscale score ranges: PCS-R: 0-16; PCS-M: 0-12; PCS-H: 0-24 A total score above 30 indicates clinically relevant level of catastrophizing
Change from baseline in the Hospital Anxiety and Depression Scale | (1) at the beginning of the treatment (T0), (2) four weeks after the end of the treatment (T3).
  The hospital anxiety and depression scale (HADS) was developed to screen for depression and anxiety in hospitalized patients. The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21).

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Çelebi University Atatürk Training and Research Hospital, Izmir, Karabaglar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhou J, Wang Y, Luo X, Fitzgerald PB, Cash RFH, Fitzgibbon BM, Che X. Revisiting the effects of rTMS over the dorsolateral prefrontal cortex on pain: An updated systematic review and meta-analysis. Brain Stimul. 2024 Jul-Aug;17(4):928-937. doi: 10.1016/j.brs.2024.07.011. Epub 2024 Jul 30. PMID 39089648
- [Result] Cheng YC, Chen WY, Su MI, Tu YK, Chiu CC, Huang WL. Efficacy of neuromodulation on the treatment of fibromyalgia: A network meta-analysis. Gen Hosp Psychiatry. 2024 Mar-Apr;87:103-123. doi: 10.1016/j.genhosppsych.2024.01.007. Epub 2024 Jan 26. PMID 38382420
- [Result] Naik A, Bah M, Govande M, Palsgaard P, Dharnipragada R, Shaffer A, Air EL, Cramer SW, Croarkin PE, Arnold PM. Optimal Frequency in Repetitive Transcranial Magnetic Stimulation for the Management of Chronic Pain: A Network Meta-Analysis of Randomized Controlled Trials. World Neurosurg. 2024 Apr;184:e53-e64. doi: 10.1016/j.wneu.2024.01.010. Epub 2024 Jan 6. PMID 38185460
- [Result] Kankane AK, Pandey AK, Ramesh PM, Agarwal A. Role of Repetitive Transcranial Magnetic Stimulation in Treatment of Fibromyalgia: A Randomized Controlled Trial. Ann Indian Acad Neurol. 2024 Mar-Apr;27(2):158-164. doi: 10.4103/aian.aian_1041_23. Epub 2024 Apr 26. PMID 38751921
- [Result] Hauser W, Ablin J, Fitzcharles MA, Littlejohn G, Luciano JV, Usui C, Walitt B. Fibromyalgia. Nat Rev Dis Primers. 2015 Aug 13;1:15022. doi: 10.1038/nrdp.2015.22. PMID 27189527
- [Result] Macfarlane GJ, Kronisch C, Dean LE, Atzeni F, Hauser W, Fluss E, Choy E, Kosek E, Amris K, Branco J, Dincer F, Leino-Arjas P, Longley K, McCarthy GM, Makri S, Perrot S, Sarzi-Puttini P, Taylor A, Jones GT. EULAR revised recommendations for the management of fibromyalgia. Ann Rheum Dis. 2017 Feb;76(2):318-328. doi: 10.1136/annrheumdis-2016-209724. Epub 2016 Jul 4. PMID 27377815
- [Result] Schweiger V, Martini A, Nizzero M, Bonora E, Del Balzo G, Gottin L, Torroni L, Polati L, Zuliani G, Secchettin E, Polati E. Prevalence of FMS Diagnosis According to ACR 2016 Revised Criteria in a Pain Therapy Centre in Italy: Observational Study. Medicina (Kaunas). 2024 Apr 4;60(4):599. doi: 10.3390/medicina60040599. PMID 38674245
- [Result] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RL, Mease PJ, Russell AS, Russell IJ, Walitt B. 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria. Semin Arthritis Rheum. 2016 Dec;46(3):319-329. doi: 10.1016/j.semarthrit.2016.08.012. Epub 2016 Aug 30. PMID 27916278
- [Result] Kaltsas G, Tsiveriotis K. Fibromyalgia. 2023 Nov 9. In: Feingold KR, Adler RA, Ahmed SF, Anawalt B, Blackman MR, Chrousos G, Corpas E, de Herder WW, Dhatariya K, Dungan K, Hamilton E, Hofland J, Jan de Beur S, Kalra S, Kaltsas G, Kapoor N, Kim M, Koch C, Kopp P, Korbonits M, Kovacs CS, Kuohung W, Laferrere B, Levy M, McGee EA, McLachlan R, Muzumdar R, Purnell J, Rey R, Sahay R, Shah AS, Sperling MA, Stratakis CA, Trence DL, Wilson DP, editors. Endotext [Internet]. South Dartmouth (MA): MDText.com, Inc.; 2000-. Available from http://www.ncbi.nlm.nih.gov/books/NBK279092/ PMID 25905317
- [Result] Perrot S, Choy E, Petersel D, Ginovker A, Kramer E. Survey of physician experiences and perceptions about the diagnosis and treatment of fibromyalgia. BMC Health Serv Res. 2012 Oct 10;12:356. doi: 10.1186/1472-6963-12-356. PMID 23051101
- [Result] Marques AP, Santo ASDE, Berssaneti AA, Matsutani LA, Yuan SLK. Prevalence of fibromyalgia: literature review update. Rev Bras Reumatol Engl Ed. 2017 Jul-Aug;57(4):356-363. doi: 10.1016/j.rbre.2017.01.005. Epub 2017 Feb 8. English, Portuguese. PMID 28743363
- [Result] Galvez-Sanchez CM, Reyes Del Paso GA. Diagnostic Criteria for Fibromyalgia: Critical Review and Future Perspectives. J Clin Med. 2020 Apr 23;9(4):1219. doi: 10.3390/jcm9041219. PMID 32340369
- [Result] Garip Y, Öztaş D, Güler T. Türk geriatrik popülasyonunda fibromiyaljinin yaygınlığı ve yaşam kalitesine etkisi. Ağrı. 2016; 28 :165-170.
- [Result] Kia S, Choy E. Update on Treatment Guideline in Fibromyalgia Syndrome with Focus on Pharmacology. Biomedicines. 2017 May 8;5(2):20. doi: 10.3390/biomedicines5020020. PMID 28536363